CLINICAL TRIAL: NCT00410696
Title: Pegfilgrastim Versus Filgrastim After High-dose Chemotherapy With Peripheral Autologous Stem Cell Reinfusion in Patients With Hematological Neoplasms and Solid Tumors: Phase II Randomised Trial
Brief Title: Pegfilgrastim Versus Filgrastim After High-dose Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Armando Santoro, MD (Other)
Responsible Party: Sponsor-Investigator, Armando Santoro, MD, MD, Istituto Clinico Humanitas
Organization: Istituto Clinico Humanitas (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ONC-2006-001; EUDRACT 2006-001409-27
Record Dates: First submitted 2006-12-12; First posted 2006-12-13 (Estimated); Last update posted 2013-07-01 (Estimated); Status verified 2013-06

CONDITIONS: Hematological Neoplasms; Tumors
Keywords: High-dose chemotherapy; Growth factor; Pegfilgrastim
MeSH Terms: conditions — Hematologic Neoplasms; Neoplasms | interventions — Filgrastim; pegfilgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Filgrastim (Active Comparator): Filgrastim administration starting 1 day after autologous stem-cell reinfusion up to hemopoietic reconstitution (defined as more than 500/mm3 for 2 days)
  Interventions: Drug: Filgrastim
- Pegfilgrastim (Experimental): Pegfilgrastim administered the day after autologous stem-cell reinfusion
  Interventions: Drug: Pegfilgrastim

INTERVENTIONS:
Drug: Filgrastim — 5 mcg/kg/day sc from day +1 after transplantation to hemopoietic reconstitution
  Other Names: Granulokine
  Arms: Filgrastim
Drug: Pegfilgrastim — 6 mg/day sc at day +1
  Other Names: Neulasta
  Arms: Pegfilgrastim

SUMMARY:
The primary objective of the study is to evaluate the efficacy and the safety of pegfilgrastim versus filgrastim, administered after high-dose chemotherapy and peripheral stem cell reinfusion.

DETAILED DESCRIPTION:
Secondary objective is to evaluate the immunological reconstitution after pegfilgrastim and filgrastim.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hematological neoplasms or solid tumors candidable to high-dose chemotherapy with autologous peripheral stem cell reinfusion
* Adequate organ function
* Written informed consent.

Exclusion Criteria:

* Use of other experimental drugs
* Active infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2006-09; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Duration of aplasia period | At time of discharge from Unit

SECONDARY OUTCOMES:
Immunological reconstitution | 1 year after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Armando Santoro, MD, Study Director — Istituto Clinico Humanitas
Locations (1):
- Istituto Clinico Humanitas, Rozzano, Milan, Italy

REFERENCES:
- [Background] Holmes FA, O'Shaughnessy JA, Vukelja S, Jones SE, Shogan J, Savin M, Glaspy J, Moore M, Meza L, Wiznitzer I, Neumann TA, Hill LR, Liang BC. Blinded, randomized, multicenter study to evaluate single administration pegfilgrastim once per cycle versus daily filgrastim as an adjunct to chemotherapy in patients with high-risk stage II or stage III/IV breast cancer. J Clin Oncol. 2002 Feb 1;20(3):727-31. doi: 10.1200/JCO.2002.20.3.727. PMID 11821454
- [Background] Farese AM, Yang BB, Roskos L, Stead RB, MacVittie TJ. Pegfilgrastim, a sustained-duration form of filgrastim, significantly improves neutrophil recovery after autologous marrow transplantation in rhesus macaques. Bone Marrow Transplant. 2003 Aug;32(4):399-404. doi: 10.1038/sj.bmt.1704156. PMID 12900776
- [Derived] Castagna L, Bramanti S, Levis A, Michieli MG, Anastasia A, Mazza R, Giordano L, Sarina B, Todisco E, Gregorini AI, Santoro A. Pegfilgrastim versus filgrastim after high-dose chemotherapy and autologous peripheral blood stem cell support. Ann Oncol. 2010 Jul;21(7):1482-1485. doi: 10.1093/annonc/mdp576. Epub 2009 Dec 11. PMID 20007996